CLINICAL TRIAL: NCT00038974
Title: Study of Viral Resistance to Antiviral Therapy of Chronic Hepatitis C (Virahep-C)
Brief Title: Hepatitis C Antiviral Resistance in African-Americans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Cancer Institute (NCI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Virahep-C (completed); U01DK060329 (NIH); U01DK060340 (NIH); U01DK060324 (NIH); U01DK060344 (NIH); U01DK060327 (NIH); U01DK060335 (NIH); U01DK060352 (NIH); U01DK060342 (NIH); U01DK060345 (NIH); U01DK060309 (NIH); U01DK060346 (NIH); U01DK060349 (NIH); U01DK060341 (NIH)
Record Dates: First submitted 2002-06-05; First posted 2002-06-10 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Interferon; Ribavirin; Efficacy; Viral load; Genetics; Cytokines; Immunology
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interferon and rivavirin (Experimental): All patients received peginterferon alfa-2a in a dose of 180 μg weekly and ribavirin in a dose of 1000 (for patients with a body weight of ⩽75 kg) or 1200 mg (for those with a body weight of >75 kg) daily.
  Interventions: Drug: peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: peginterferon alfa-2a
Drug: Ribavirin

SUMMARY:
This study is designed to test the hypothesis that African-Americans respond less well to combination pegylated interferon and ribavirin therapy than Caucasian-Americans who have chronic hepatitis C genotype 1 and who were not previously treated with either interferon or ribavirin. Reasons for differences in response, regardless of race, will be studied.

ELIGIBILITY:
Inclusion:

* Age between 18 and 70 years at screening
* Black/African American or White/Caucasian
* Born in the United States
* Quantifiable Serum HCV RNA
* Hepatitis C genotype 1
* Liver biopsy consistent with chronic hepatitis C
* Negative urine pregnancy test
* Males and Females must be using two reliable forms of effective contraception while on drug and during follow-up.

Exclusion:

* Previous treatment with interferon or ribavirin
* Positive test at screening for anti-HIV
* Positive test for HBsAg
* Alcohol consumption of more than two drinks/day
* History of other chronic liver disease
* Pregnant or breast-feeding women
* Male partners of women who are pregnant or contemplating pregnancy
* Neutrophil count <1000 cells/mm3
* Hgb <11 g/dl in women or 12 g/dl in men
* Platelet count <75,000 cells/mm3.
* Thalassemia, spherocytosis, history of GI bleeding or those at increased risk of anemia
* Serum creatinine level >1.5 times the upper limit of normal at screening or CrCl < 75cc/min
* Current dialysis
* Alcohol or drug abuse within 6 months
* Current (<6 months)severe psychiatric disorder
* History of immunologically mediated disease
* Decompensated liver disease
* High risk cardiovascular/coronary artery disease
* Severe seizure disorder or anticonvulsant use
* Solid organ or bone marrow transplantation
* Thyroid disease poorly controlled on prescribed medications
* History or other evidence of retinopathy
* Chronic use of oral steroids
* Inability or unwillingness to provide informed consent or abide by the study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2002-08; Primary Completion 2004-12 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response (SVR) | 24 weeks after therapy is discontinued
  The primary end point of therapy was an SVR that was definied as the absences of detectable HCV RNA in serum 24 weeks after therapy was stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Robuck, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - University of Miami School of Medicine, Miami, Florida
  - Rush University, Chicago, Illinois
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - New York-Presbyterian Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available in the NIDDK Central Repository
Supporting Information: Study Protocol, ICF, CSR
URL: https://www.niddkrepository.org/search/study/?q=virahep+c

REFERENCES:
- [Result] Conjeevaram HS, Fried MW, Jeffers LJ, Terrault NA, Wiley-Lucas TE, Afdhal N, Brown RS, Belle SH, Hoofnagle JH, Kleiner DE, Howell CD; Virahep-C Study Group. Peginterferon and ribavirin treatment in African American and Caucasian American patients with hepatitis C genotype 1. Gastroenterology. 2006 Aug;131(2):470-7. doi: 10.1053/j.gastro.2006.06.008. PMID 16890601
- [Derived] Sarkar S, Jiang Z, Evon DM, Wahed AS, Hoofnagle JH. Fatigue before, during and after antiviral therapy of chronic hepatitis C: results from the Virahep-C study. J Hepatol. 2012 Nov;57(5):946-52. doi: 10.1016/j.jhep.2012.06.030. Epub 2012 Jul 1. PMID 22760009
- [Derived] Dove LM, Rosen RC, Ramcharran D, Wahed AS, Belle SH, Brown RS, Hoofnagle JH; Virahep-C Study Group. Decline in male sexual desire, function, and satisfaction during and after antiviral therapy for chronic hepatitis C. Gastroenterology. 2009 Sep;137(3):873-84, 884.e1. doi: 10.1053/j.gastro.2009.05.060. Epub 2009 Jun 13. PMID 19527724
- [Derived] Hoofnagle JH, Wahed AS, Brown RS Jr, Howell CD, Belle SH; Virahep-C Study Group. Early changes in hepatitis C virus (HCV) levels in response to peginterferon and ribavirin treatment in patients with chronic HCV genotype 1 infection. J Infect Dis. 2009 Apr 15;199(8):1112-20. doi: 10.1086/597384. PMID 19284286
- [Derived] Cannon NA, Donlin MJ, Fan X, Aurora R, Tavis JE; Virahep-C Study Group. Hepatitis C virus diversity and evolution in the full open-reading frame during antiviral therapy. PLoS One. 2008 May 7;3(5):e2123. doi: 10.1371/journal.pone.0002123. PMID 18463735